CLINICAL TRIAL: NCT01139216
Title: Effect of DAIKENCHUTO (TU-100), a Gastrointestinal Nerve Modulator, on Rectal Compliance, Rectal Sensation and Small Bowel and Colonic Transit in Female Patients With Functional Constipation
Brief Title: Effect of TU-100 on Rectal Compliance, Rectal Sensation and Small Bowel and Colonic Transit in Females With Constipation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Tsumura USA (Industry)
Collaborators: Cato Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TU100CPT2
Record Dates: First submitted 2010-06-03; First posted 2010-06-08 (Estimated); Last update posted 2013-01-14 (Estimated); Status verified 2013-01

CONDITIONS: Functional Constipation; Gastric Emptying; Whole Gut Transit; Small Bowel Transit; Colonic Transit; Rectal Compliance; Rectal Sensation
Keywords: Digestive system diseases; Gastrointestinal diseases; Intestinal diseases; Colonic inertia
MeSH Terms: conditions — Digestive System Diseases; Gastrointestinal Diseases; Intestinal Diseases; Constipation | interventions — dai-kenchu-to; 12,13-dihydro-N-methyl-6,11,13-trioxo-5H-benzo(4,5)cyclohepta(1,2-b)naphthalen-5,12-imine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Daikenchuto (TU-100) 7.5g/day (Experimental): Daikenchuto (TU-100) 2.5g TID (7.5g/day)
  Interventions: Drug: Daikenchuto (TU-100)
- Daikenchuto (TU-100) 15g/day (Experimental): Daikenchuto (TU-100) 5g TID (15g/day)
  Interventions: Drug: Daikenchuto (TU-100)
- Placebo (Placebo Comparator): Placebo TID
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Daikenchuto (TU-100) — Subjects will receive 2.5g TID (7.5g/day) of TU-100. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 4 weeks.
  Arms: Daikenchuto (TU-100) 7.5g/day
Drug: Daikenchuto (TU-100) — Subjects will receive 5g TID (15g/day) of TU-100. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 4 weeks.
  Arms: Daikenchuto (TU-100) 15g/day
Drug: Placebo — Subjects will receive daily dose of TU-100 placebo. Dosage form is granule. Subject will take a daily dose divided 3 times per day for 4 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the dose-related effects of TU-100, a botanical agent that modulates gastrointestinal nerves, on rectal compliance, rectal sensation thresholds and small bowel and colonic transit in female patients with functional constipation as compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Meet Rome III criteria for functional constipation
2. Willing and able to provide written informed consent
3. Females, not pregnant or not breast-feeding

   * Females of childbearing potential must use an acceptable form of contraception during the study and for 30 days after the last dose. Acceptable methods include surgical sterilization, hormonal contraceptives (such as oral contraceptives, Depo-Provera, Nuva Ring, condoms used with a spermicide, an IUD or abstinence.
   * Females are not considered to be of childbearing potential if they are postmenopausal for at least two years or have been surgically sterilized.
4. Ages 18 to 65 years old inclusive
5. A body mass index (BMI) between 18 and 40 kg/m2 inclusive
6. A negative urine drug screen at Visit 1
7. Normal or not clinically significant laboratory results as reviewed by the study physicians
8. A normal rectal exam result on file within the past 2 years or performed at Visit 1 in order to exclude the possibility of an evacuation disorder. Examination must exclude findings suggestive of an evacuation disorder such as high sphincter tone at rest, failure of perineal descent and spasm, tenderness or paradoxical contraction of the puborectalis muscles.
9. Do not have sufficient criteria for irritable bowel syndrome (IBS)

Exclusion Criteria:

1. Structural or metabolic diseases/conditions that affect the gastrointestinal system or functional gastrointestinal disorders other than constipation.
2. Taking any medication that in the opinion of the principal investigator has a potential to alter GI transit. This includes but is not limited to osmotic or stimulant laxatives, magnesium or aluminum-containing antacids, prokinetics, erythromycin, narcotics, anticholinergics, selective norepinephrine reuptake inhibitors (SNRIs), opiates, GABAergic agents and benzodiazepines.

   * Note: Tricyclic antidepressants are permissible at doses equal to or less than 25 mg daily; selective serotonin reuptake inhibitor (SSRI) antidepressants are permissible at low, stable doses. Analgesics such as Tylenol, ibuprofen, naproxen and aspirin are permissible. All medications shall be reviewed by the principal investigator on a case by case basis.
   * Rescue medications: Rescue medications shall be reviewed and approved as necessary for exacerbation of constipation as the study medication treatment period is lengthy, about 28 days total. The patient will contact the study staff to request review and approval of the use of a rescue medication by the principal investigator. The use of the rescue medication will be documented by the patient in the bowel pattern diary. Rescue medications are not allowed within 7 days of the abbreviated baseline or the full transit scintigraphy to ensure data integrity.
3. Clinical evidence, including but not limited to a clinically significant abnormal physical exam or laboratory test result or a past event documented in the past medical record, or current clinically significant abnormal physical exam or laboratory test result that could indicate significant cardiovascular, respiratory, renal, hepatic, gastrointestinal, hematological, neurological, psychiatric or other diseases that interfere with the objectives of the study. If a laboratory test result is abnormal and clinically significant, it may be repeated once at the discretion of the principal investigator. If the laboratory test result remains abnormal and clinically significant, the patient will be discontinued from the study and referred to a primary care physician for evaluation.
4. Patients who are considered to be alcoholics not in remission or known substance abusers.
5. Patients who have participated in another clinical study in the past 30 days.
6. Patients who have a history of allergic reactions to egg, ginseng, ginger or Sichuan pepper
7. Patients who are clinically lactose intolerant
8. Patients must agree to avoid alcohol during the days of Visits 5, 6 and 7 to avoid corrupting the data from the anorectal manometry and rectal barostat tests.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Colonic geometric center at 24 hours measured by scintigraphy | Up to 48 hours
T1/2 of ascending colon emptying as measured by scintigraphy | Up to 48 hours

SECONDARY OUTCOMES:
Colonic geometric center at 4 hours and 48 hours | Up to 48 hours
Colonic filling at 6 hours | Up to 48 hours
t1/2 of gastric emptying of solid | Up to 48 hours
Rectal Compliance Pr1/2 | Up to 3 hours
Rectal sensation thresholds (gas, urgency to defecate, and pain) | Up to 3 hours
Anal sphincter pressure at rest | Up to 3 hours
Anal sphincter pressure during squeeze | Up to 3 hours
Recto-anal pressure difference during straining to simulate defecation | Up to 3 hours
Stool frequency | 6 weeks
Stool consistency | 6 weeks
PAC-QOL (Patient Assessment of Constipation Quality of Life) score | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester Methodist CRU, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Iturrino J, Camilleri M, Wong BS, Linker Nord SJ, Burton D, Zinsmeister AR. Randomised clinical trial: the effects of daikenchuto, TU-100, on gastrointestinal and colonic transit, anorectal and bowel function in female patients with functional constipation. Aliment Pharmacol Ther. 2013 Apr;37(8):776-85. doi: 10.1111/apt.12264. Epub 2013 Mar 4. PMID 23451764